CLINICAL TRIAL: NCT06773520
Title: Use of Three-dimensional Transvaginal Ultrasound for Anal Sphincter Evaluation: "A New Technique"
Brief Title: Use of Three-dimensional Transvaginal Ultrasound for Anal Sphincter Evaluation
Acronym: 3D_TV_OASIS
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: 3D_TV_OASIS
Record Dates: First submitted 2024-12-03; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-10

CONDITIONS: Obstetric Anal Sphincter Injury
Keywords: 3D untrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the reproducibility of new 3D/4D ultrasound volume analysis techniques in the assessment of anal sphincter integrity and thickness in both pregnancy and immediate postpartum.

The negative impact that OASISs (Obstetric Anal Sphincter Injuries), and possible subsequent anal incontinence, have on women's quality of life has stimulated research in this field in recent decades. However, there are still few studies concerning the topic. The transperineal approach by means of the transvaginal probe in the study of the pelvic floor, anal sphincter and related lesions has helped us to make strides in our knowledge of the anatomy of the pelvic floor and in defining the lesions that may affect it.

DETAILED DESCRIPTION:
The development of ultrasound techniques such as 3D and 4D and new reproducible and increasingly accurate volumetric acquisition modalities shows promise for improving the diagnosis of OASIS and the clinical management of OASIS and consequently the quality of life of women.

With new, simpler techniques of 3D/4D volume analysis of the anal sphincter, the number of operators able to objectively and accurately assess anal sphincter integrity, both in the delivery room and postpartum, could increase. The application and dissemination of an accurate and reproducible technique in the subjective assessment of the anal sphincter could help operators improve and refine the technique of surgical correction of anal sphincter injuries.

The primary objective of the study is to evaluate the reproducibility of novel 3D/4D ultrasound volume analysis techniques, using curvilinear reconstruction of the coronal plane of the anal sphincter combined with contrast enhancement technique (optic OMNIVIEW), in the assessment of anal sphincter integrity and thickness, both in pregnancy and immediate postpartum.

Secondary objectives include:

* Evaluation of the feasibility of new off-line analysis techniques.
* Evaluation of the correlation between thickness and ultrasound integrity of the anal sphincter at the postpartum visit and women's symptomatology in the postpartum.

To reduce bias as much as possible, each operator during each assessment will be "blinded" to the patient's history and all other measurements.

Clinicians who perform more than one measurement per volume will do so at least one month apart between each measurement.

The patient will be treated according to common clinical practice ensuring the standard of care. Patients will not undertake additional visits to those routinely performed. This is an evaluation of new techniques for off-line (in the absence of the patient) analysis of ultrasound volumes that are currently part of routine visits in both pre and postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant nulliparous or primiparous women;
* Age between 18 and 44 years
* Acquisition of informed consent form

Exclusion Criteria:

None

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Nulliparous and primiparous pregnant women. Participants will be enrolled at the Division of Obstetrics and Prenatal Age Medicine (IRCCS - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola). Participants will be enrolled during the obstetrical visit or during hospitalization or during visits in the postpartum period.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Intraclass correlation coefficient (ICC) | At the end of pregnancy (up to 40 weeks of gestation)
  Bland-Altman analysis
Presence of a systematic difference between the various measures taken by different operators | At the end of pregnancy (up to 40 weeks of gestation)
  Bland-Altman analysis
Dispersion of the differences between the measures taken by two different operators and the two measures taken by the same operator around the mean of the respective differences. | At the end of pregnancy (up to 40 weeks of gestation)
  Bland-Altman analysis

SECONDARY OUTCOMES:
Percentage of volumes acquired in which measurement of the external anal sphincter will be feasible | At the end of pregnancy (up to 40 weeks of gestation)
  New analysis techniques: curvilinear reconstruction of the coronal plane of the anal sphincter combined with contrast enhancement technique.
Correlation between anal sphincter thickness and the presence of symptoms related to rectal incontinence | At the end of pregnancy (up to 40 weeks of gestation)
  Comparison of anal sphincter thickness between women with and without exintent signs of rectal incontinence at postpartum visit

CONTACTS AND LOCATIONS:
Overall Officials: Aly Mohamed Alaaeldin Kamaleldin Aly Youssef, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy